CLINICAL TRIAL: NCT02371317
Title: Stress Management for High Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kent State University (Other)
Collaborators: University of Pennsylvania (Other); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, David M. Fresco, Professor, Kent State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: KentSU
Record Dates: First submitted 2015-01-21; First posted 2015-02-25 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Prehypertension
Keywords: Randomized clinical trial; Early medical intervention; Intervention studies; Blood pressure; Stress Management
MeSH Terms: conditions — Prehypertension | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mindfulness-Based Stress Reduction (Experimental): The Mindfulness-Based Stress Reduction intervention includes eight 2.5-hour weekly group sessions and an all-day retreat.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction; Other: American Heart Association Recommended Self-Care
- Stress Management Education (Active Comparator): The Stress Management Education intervention includes eight 2.5-hour weekly group sessions and an all-day retreat.
  Interventions: Behavioral: Stress Management Education; Other: American Heart Association Recommended Self-Care
- AHA Recommended Self-Care (Other): All participants will receive the American Heart Association - Understanding and Controlling Your High Blood Pressure Brochure and information on the Dietary Approach to Stop Hypertension from the National Institutes of Health. These brochures describe ways that individuals can improve their lifestyle through better diet and exercise. Participants will get a chance to try and make healthy lifestyle changes on their own, using this information.
  Interventions: Other: American Heart Association Recommended Self-Care

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — Patients are randomized to an intervention
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Stress Management Education — Patients are randomized to an intervention
  Other Names: SME
  Arms: Stress Management Education
Other: American Heart Association Recommended Self-Care — All Patients receive AHA Recommended Self-Care

SUMMARY:
The purpose of this research study is to examine the efficacy of two stress management interventions in reducing blood pressure (BP) in patients who have prehypertension (BP between 120/80 and 139/89). It is expected that participants will be better able to control their BP through reducing stress and increasing healthy lifestyle behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Unmedicated high blood pressure (SBP of 120-139 or DBP of 80-89)
* BMI in the range of 19-40
* Interest in attempting to control blood pressure through lifestyle modification

Exclusion Criteria:

* pacemakers
* uncontrolled hypertension (SBP≥140 or DBP≥90)
* atrial fibrillation
* myocardial infarction (MI)
* percutaneous transluminal coronary angioplasty (PTCA)
* coronary artery bypass graft (CABG) within 6 months of enrollment
* congestive heart failure
* uncorrected primary valvular disease hypertrophic or restrictive cardiomyopathy
* uncorrected thyroid heart disease
* chronic kidney disease
* persistent tachyarrhythmia
* JNC risk category C (target organ damage, diabetes)
* patients who are pregnant or plan to become pregnant within 9 months
* patients who are lactating
* patients unable to comply with assessment procedures
* patients with alcohol or drug abuse within 12 months
* patients who consume more than 21 alcoholic drinks per week
* patients who are current smokers
* patients who are unable to provide informed consent or who have dementia
* patients with previous extensive meditation or yoga training
* patients with blood pressure ≥140/90

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Clinic Blood Pressure | Week 0, Week 4, Week 8, Week 34, and Week 60
  All clinic blood pressure assessments will be completed in a quiet, climate controlled room according to American Heart Association guidelines. The mean of the three seated readings on the non- dominant arm will be averaged to define clinic blood pressure.
Change in Diastolic Clinic Blood Pressure | Week 0, Week 4, Week 8, Week 34, and Week 60
  All clinic blood pressure assessments will be completed in a quiet, climate controlled room according to American Heart Association guidelines. The mean of the three seated readings on the non- dominant arm will be averaged to define clinic blood pressure.

SECONDARY OUTCOMES:
Change in 24-hour Ambulatory Systolic Blood Pressure | Week 0, Week 8, Week 60
  Participants will complete 24-hour Ambulatory Blood Pressure Monitoring with the Oscar 2 oscillometric blood pressure monitor. The Oscar will be programmed to take three blood pressure measurements per hour from 6 AM till 11 PM and two BP measurements per hour from 11 PM to 6 AM. During each reading, participants will be instructed to drop their arms to their sides as soon as they sense the cuff inflating, and to keep it relaxed and still until a few seconds after the deflation has finished. Ambulatory SBP and DBP will be derived by computing the mean of all valid readings obtained during waking hours and nighttime sleep.
Change in 24-hour Ambulatory Diastolic Blood Pressure | Week 0, Week 8, Week 60
  Participants will complete 24-hour Ambulatory Blood Pressure Monitoring with the Oscar 2 oscillometric blood pressure monitor. The Oscar will be programmed to take three blood pressure measurements per hour from 6 AM till 11 PM and two BP measurements per hour from 11 PM to 6 AM. During each reading, participants will be instructed to drop their arms to their sides as soon as they sense the cuff inflating, and to keep it relaxed and still until a few seconds after the deflation has finished. Ambulatory SBP and DBP will be derived by computing the mean of all valid readings obtained during waking hours and nighttime sleep.

CONTACTS AND LOCATIONS:
Overall Officials: David M Fresco, Ph.D., Principal Investigator — Kent State University
Locations (2):
- United States (2):
  - W.O. Walker Building, Cleveland, Ohio
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Hughes JW, Fresco DM, Myerscough R, van Dulmen MH, Carlson LE, Josephson R. Randomized controlled trial of mindfulness-based stress reduction for prehypertension. Psychosom Med. 2013 Oct;75(8):721-8. doi: 10.1097/PSY.0b013e3182a3e4e5. PMID 24127622
- [Derived] Chin GR, Greeson JM, Hughes JW, Fresco DM. Does Dispositional Mindfulness Predict Cardiovascular Reactivity to Emotional Stress in Prehypertension? Latent Growth Curve Analyses from the Serenity Study. Mindfulness (N Y). 2021 Nov;12(11):2624-2634. doi: 10.1007/s12671-021-01745-y. Epub 2021 Sep 18. PMID 35694435